CLINICAL TRIAL: NCT06916689
Title: Efficacy And Tolerability Of The Asymmetric Split Regimen With A Very Low Volume Bowel Preparation: Split-The-Split Study
Brief Title: Efficacy And Tolerability Of Asymmetric Split Regimen For Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Rhodense (Other)
Responsible Party: Principal Investigator, gianpiero manes, Head of the Gastroenterology Unit, ASST Rhodense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 101-17022023
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2023-03

CONDITIONS: Colon Preparation; Polyps Colorectal
Keywords: Asymmetric split regimen; Bowel preparation; Colon cleansing; Very low volume preparation; 1L PEG + ascorbate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Asymmetric split dose preparation (Experimental): 75% of the dose is given on the day before of the procedure and 25% of the dose is given on the day of the procedure
  Interventions: Drug: 1L PEG-Asc
- Symmetric split dose preparation (Active Comparator): 50% of the dose is given on the day before of the procedure and 50% of the dose is given on the day of the procedure
  Interventions: Drug: 1L PEG-Asc

INTERVENTIONS:
Drug: 1L PEG-Asc — PEG 3350 plus sodium sulfate plus sodium chloride plus potassium chloride plus ascorbic acid plus sodium ascorbate

SUMMARY:
The investigators aimed to compare the efficacy for bowel cleansing of a split-dose regimen with a low morning dose of PEG solution (Asymmetric; 25% of the dose is given on the day of the procedure and 75% of the dose is given on the day before) with the standard split-dose regimen in patients undergoing screening and surveillance colonoscopy using a very low volume bowel preparation (1L PEG+Ascorbate). Consecutive outpatients undergoing screening and surveillance colonoscopy were enrolled in a randomized, single-blind, non-inferiority clinical trial. Patients were randomly assigned to: group A, asymmetric split dose regimen (0,75 L of PEG + ASC the day before and 0,25 L 2:30 hours before colonoscopy); group B, symmetric split dose regimen (0,5 L of PEG + ASC the day before and 0,5 L 3 hours before colonoscopy). Primary endpoint was the proportion of adequate bowel cleansing. Moreover, all patients filled in a validated, nurse-administered questionnaire assessing compliance, tolerability and safety of bowel preparation.

DETAILED DESCRIPTION:
Prospective observational, single-blind study conducted in two endoscopy centers belonging to the same Local Health Authority. The two bowel preparation regimens under study (symmetric split and asymmetric split) will be compared in a population of patients undergoing screening for colorectal cancer.

Patient enrollment, product prescription, and the subsequent pre-endoscopic evaluation of safety, tolerability, acceptability, and compliance will be carried out by an assistant who will not be blinded to the type of preparation used.

Endoscopic evaluation, however, will be performed by an experienced endoscopist who will be blinded to the type of bowel preparation administered to the patient.

The bowel preparation product used consists of a very low-volume solution of Macrogol (3350) + Ascorbic Acid (1 liter) (PLENVU®, Norgine).

Bowel cleanliness level assessed using the Boston Bowel Preparation Scale adn overall tolerability of bowel preparation are primary outcomes.

Patient compliance and safety; the number of detected lesions, the percentage of complete colonoscopies, the duration of the colonoscopy, the degree of discomfort/pain perceived by the patient during the examination, and procedure-related complications are secondary outcomes.

Patients will be assigned to the two treatment groups according to a computer-generated sequence.

Data will be expressed as mean and standard deviation for quantitative variables and as frequencies for qualitative variables. The comparison between the two groups will be performed using the t-test for quantitative variables and the chi-square (χ²) test for qualitative variables.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled as outpatient for screening or surveillance colonoscopy

Exclusion Criteria:

* Inpatients
* refusal of split dose regimen for bowel preparation
* previous history of colorectal resection
* severe cardiac disease
* advanced (stage IV and V) chronic kidney disease
* pregnancy; ileus
* suspected bowel obstruction or toxic megacolon
* known inflammatory bowel disease
* known or suspected allergy to PEG.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Quality of bowel prepreparation | 2 days
  Quality of bowel prepreparation/cleanliness scored using the Boston Bowel Preparation Scale. Each segment of the colon received a score from 0 to 3, and these segment scores were summed for a total BBPS score ranging from 0 to 9. The preparation was considered adequate when BBPS score was ≥ 6 with a score with at least 2 points in any segment

SECONDARY OUTCOMES:
Adenoma detection rate | 2 days
  rate of patients with at least one adenoma
Rate of the occurrence of adverse events | 2 days
  Rate of the occurrence of adverse events (bad taste in mouth, gastric fullness, nausea or vomiting, bloating, abdominal pain, headache)
Compliance | 2 days
  Compliance was assessed by the amount of intake of study agents using a 3-point scale: 1 (100% intake), 2 (≥ 75% intake), and 3 (< 75% intake).
Tolerability of the preparation, as reported by the patient on a Validated Questionnaire | 2 days
  Tolerability was evaluated assessing how patient finds tolerable the bowel preparation by using a 4-point scale: 1 (Easy), 2 (Acceptable), 3 (Somewhat difficult), 4 (Very difficult), plus a Visual Scale with a number from 0 (untolerable) to 100 (very tolerable).

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiero Manes, Principal Investigator — ASST Rhodense
Locations (1):
- ASST Rhodense, Garbagnate Milanese, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided